CLINICAL TRIAL: NCT06568848
Title: Effects of EKKO Versus Conservative Treatment for Gross Motor Functions in Cerebral Palsy Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/739
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exp Group (Experimental)
  Interventions: Combination Product: EKKO therapy
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: Conservative Treatment

INTERVENTIONS:
Combination Product: EKKO therapy — In this group 6 particepents will be included .the interventions will be given for 10 seconds on each finger tips . the session will be 30 mins. 4 to 5 sessions per week
  Arms: Exp Group
Diagnostic Test: Conservative Treatment — In this group 6 participants will be included .: Conservative treatment, which includes ROM isometric exercises (20 repetitions per limb), stretching exercises (10 seconds per limb with 3 repetitions), balance training (standing without belts for 20 minutes), and gait training (walking with a frame). The session will be 30 mins
  Arms: Control Group

SUMMARY:
"Cerebral palsy (CP) affects gross motor function variably, with the spastic type notably impacting movement, coordination, and balance. Research highlights that spastic CP, characterized by muscle stiffness, can severely hinder activities like walking and running. Interventions such as gait training and vibrational therapy have shown promise in enhancing muscle function and body movements. A new device, EKKO, uses vibrational waves based on Neurotransmission Cognitive Theory to improve gross motor skills in children with CP by applying mechanical vibrations to nerve points.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of EKKO therapy with traditional conservative treatments (such as range of motion exercises and balance training) in improving gross motor function in children with CP. Conducted over six months with randomized controlled trials, the research seeks to provide evidence-based insights into optimizing rehabilitation strategies for better motor performance and quality of life for CP patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. cerebral palsy (CP)
* Severity: Typically applied to those with mild to moderate CP

Exclusion Criteria:

* Participants without a confirmed diagnosis of cerebral palsy or any other neurological condition
* Severe cp cases may be excluded

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
GMFM Scale | 12 Months
  improvement in gross motor function, measured using the GMFM scale. The scale evaluates various dimensions such as sitting, rolling, jumping, crawling, kneeling, walking, and running. Assessments will be conducted at three points: pre-evaluation (month 1), mid-evaluation (month 3), and post-evaluation (end of month 6).

CONTACTS AND LOCATIONS:
Locations (1):
- Little angles home sailkot cantt aziz bhati shaheed road opposit junior aps, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No